CLINICAL TRIAL: NCT03610490
Title: Clinical Study to Assess Efficacy and Safety of MDA-TIL (Autologous Expanded Tumor Infiltrating Lymphocytes) Across Multiple Tumor Types
Brief Title: Autologous Tumor Infiltrating Lymphocytes MDA-TIL in Treating Patients With Recurrent or Refractory Ovarian Cancer, Colorectal Cancer, or Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Iovance Biotherapeutics (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0671; NCI-2018-01509 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0671 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Malignant Solid Neoplasm; Metastatic Colorectal Adenocarcinoma; Metastatic Ovarian Carcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Platinum-Resistant Ovarian Carcinoma; Recurrent High Grade Ovarian Serous Adenocarcinoma; Recurrent Ovarian Carcinosarcoma; Refractory Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Ovarian Neoplasms; Colorectal Neoplasms | interventions — Cyclophosphamide; fludarabine; Interleukin-2; 4-toluenesulfonyl fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (autologous tumor infiltrating lymphocytes MDA-TIL) (Experimental): LYMPHODEPLETION REGIMEN: Patients receive cyclophosphamide IV over 2 hours on days -7 and -6, and fludarabine IV over 15-30 minutes on days -5 to -1 in the absence of disease progression or unacceptable toxicity.
  T-CELL INFUSION: Patients receive autologous tumor infiltrating lymphocytes MDA-TIL IV over 45 minutes on day 0. Patients then receive IL-2 IV over 30 minutes on days 1-4 for up to 6 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Autologous Tumor Infiltrating Lymphocytes MDA-TIL; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Interleukin-2; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Autologous Tumor Infiltrating Lymphocytes MDA-TIL — Given IV
  Other Names: MDA Autologous TILs; MDA Autologous Tumor Infiltrating Lymphocytes; MDA-TILs
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Interleukin-2 — Given IV
  Other Names: Epidermal Thymocyte Activating Factor; ETAF; IL-2; IL2; IL2 Protein; Interleukin 2; Interleukin 2 Precursor; Interleukin II; Lymphocyte Mitogenic Factor; Mitogenic Factor; Ro-236019; T Cell Growth Factor; T-Cell Growth Factor; TCGF; Thymocyte Stimulating Factor; TSF
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well autologous tumor infiltrating lymphocytes MDA-TIL works in treating patients with ovarian cancer, colorectal cancer, or pancreatic ductal adenocarcinoma that has come back (recurrent) or does not respond to treatment (refractory). Autologous tumor infiltrating lymphocytes MDA-TIL, made by collecting and growing specialized white blood cells (called T-cells) from a patient's tumor, may help to stimulate the immune system in different ways to stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate efficacy using objective response rate (ORR) using the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 in subjects with ovarian cancer, pancreatic ductal adenocarcinoma (PDAC), and colorectal cancers.

SECONDARY OBJECTIVES:

I. Determine the disease control rate (DCR) within and across cohorts. II. Determine the duration of response (DOR). III. Determine progression-free survival (PFS) and overall survival (OS). IV. Further characterize the safety profile of adoptive cell therapy (ACT) with tumor-infiltrating lymphocytes (TIL) across multiple tumor types.

EXPLORATORY OBJECTIVES:

I. Establish duration of TIL persistence. II. Compare the molecular and immunological features of tumors before and after TIL therapy.

III. Prospectively evaluate the existing immunotherapy response criteria (immune-related Response Evaluation Criteria in Solid Tumors [irRECIST]) as the best response assessment tool for TIL therapy among a diverse group of solid tumors.

IV. Investigate TIL attributes (CD8 %, CD27 and CD28 expression) and correlation with response to therapy.

V. Assess tumor marker (CA19-9; CA-125) response in patients who produce this tumor marker.

VI. Assess Health-Related Quality of Life (HRQOL).

OUTLINE:

LYMPHODEPLETION REGIMEN: Patients receive cyclophosphamide intravenously (IV) over 2 hours on days -7 and -6, and fludarabine IV over 15-30 minutes on days -5 to -1 in the absence of disease progression or unacceptable toxicity.

T-CELL INFUSION: Patients receive autologous tumor infiltrating lymphocytes MDA-TIL IV over 45 minutes on day 0. Patients then receive IL-2 IV over 30 minutes on days 1-4 for up to 6 doses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at week 18, at 6, 9, 12, 18, and 24 months, and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide informed consent
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1 at enrollment and within 7 days of initiating lymphodepleting chemotherapy
* Subjects must have an area of tumor amenable to excisional biopsy (core biopsies may be allowed) for the generation of TIL separate from, and in addition to, a target lesion to be used for response assessment
* Any prior therapy directed at the malignant tumor, including radiation therapy, chemotherapy, and biologic/targeted agents must be discontinued at least 28 days prior to tumor resection for preparing TIL therapy
* Absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days of enrollment)
* Hemoglobin >= 9.0 g/dL (transfusion allowed) (within 7 days of enrollment)
* Platelet count >= 100,000/mm^3 (within 7 days of enrollment)
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) and aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) < 2.5 x the upper limit of normal (ULN)

  * Patients with liver metastases may have liver function test [LFT] =< 5.0 x ULN (within 7 days of enrollment)
* Calculated creatinine clearance (Cockcroft-Gault) >= 50.0 mL/min (within 7 days of enrollment)
* Total bilirubin =< 1.5 x ULN (within 7 days of enrollment)
* Prothrombin time (PT) & activated partial thromboplastin time (aPTT) =< 1.5 x ULN (correction with vitamin K allowed) unless subject is receiving anticoagulant therapy (which should be managed according to institutional norms prior to and after excisional biopsy) (within 7 days of enrollment)
* Negative serum pregnancy test (female subjects of childbearing potential) (within 7 days of enrollment)
* Subjects must not have a confirmed human immunodeficiency virus (HIV) infection
* Subjects must have a 12-lead electrocardiogram (EKG) showing no active ischemia and Fridericia's corrected QT interval (QTcF) less than 480 ms
* Subjects must also have a negative dobutamine stress echocardiogram before beginning treatment
* Subjects of childbearing potential must be willing to practice an approved highly effective method of birth control starting at the time of informed consent and for 1 year after the completion of the lymphodepletion regimen. Approved methods of birth control are as follows: hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation or hysterectomy; subject/partner status post vasectomy; implantable or injectable contraceptives; and condoms plus spermicide
* Able to adhere to the study visit schedule and other protocol requirements
* Pulmonary function tests (spirometry) demonstrating forced expiratory value (FEV) 1 greater than 65% predicted or forced vital capacity (FVC) greater than 65% of predicted
* Ovarian cancer cohort only: Subjects must have high grade non-mucinous histology (carcinosarcomas are allowed)
* Ovarian cancer cohort only: Subjects must have failed at least two prior lines of chemotherapy (i.e. frontline adjuvant chemotherapy plus one additional line for recurrent/progressive disease), or have platinum resistant disease
* Colorectal cohort only: Subjects with colorectal adenocarcinoma must have metastatic disease that is considered incurable with currently available therapies and have derived maximal benefit from or have become refractory to frontline conventional therapy (e.g. leucovorin calcium [calcium folinate], 5-fluorouracil and oxaliplatin [FOLFOX], leucovorin calcium, 5-fluorouracil, and irinotecan [FOLFIRI]).
* Colorectal cohort only: Subjects should have low disease burden such that in the treating physician's opinion the patient would not require additional intervening treatment for 7-8 weeks (required for TIL harvest and manufacturing)
* Pancreatic adenocarcinoma cohort only: Subjects must have histologically or cytologically documented diagnosis of PDAC with oligo-metastatic disease
* Pancreatic adenocarcinoma cohort only: Subjects must have progressed on, or received maximal benefit from, front-line therapy
* Pancreatic adenocarcinoma cohort only: Patients may have received unlimited lines of prior standard of care therapy
* Pancreatic adenocarcinoma cohort only: Patients with ascites or carcinomatosis are not eligible for the study
* Pancreatic adenocarcinoma cohort only: Patients will need an albumin of >= 3.0 mg/dL within 7 days of enrollment
* TREATMENT INCLUSION CRITERION: Within 24 h of starting lymphodepleting chemotherapy, subjects must meet the following laboratory criteria:

  * Absolute neutrophil count (ANC) >= 1000/mm^3
  * Hemoglobin >= 9.0 g/dL (transfusion allowed)
  * Platelet count >= 100,000/mm3
  * ALT/SGPT and AST/SGOT =< 2.5 x the upper limit of normal (ULN)

    * Patients with liver metastases may have liver function tests (LFT) =< 5.0 x ULN
  * Calculated creatinine clearance (Cockcroft-Gault) >= 50.0 mL/min
  * Total bilirubin =< 1.5 X ULN

Exclusion Criteria:

* Active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system. Principal investigator (PI) or his/her designee shall make the final determination regarding appropriateness of enrollment
* Patients with active viral hepatitis
* Patients who have a left ventricular ejection fraction (LVEF) < 45% at screening
* Patients with a history of prior adoptive cell therapies
* Persistent prior therapy-related toxicities greater than grade 2 according to Common Toxicity Criteria for Adverse Events (CTCAE) v. 4.03, except for peripheral neuropathy, alopecia, or vitiligo prior to enrollment
* Primary immunodeficiency
* History of organ or hematopoietic stem cell transplant
* Chronic steroid therapy, however prednisone or its equivalent is allowed at < 10 mg/day
* Patients who are pregnant or nursing
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his/her designee, would prevent adequate informed consent
* History of clinically significant autoimmune disease including active, known, or suspected autoimmune disease. Subjects with resolved side effects from prior checkpoint inhibitor therapy, vitiligo, psoriasis, type 1 diabetes or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded
* History of clinically significant chronic obstructive pulmonary disease (COPD), asthma, or other chronic lung disease
* History of a second malignancy (diagnosed in the last 5 years). Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* History of known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to initiation of lymphodepletion
* Has received a live vaccine within 30 days prior to the initiation of lymphodepletion
* Patients who have a contraindication to or history of hypersensitivity reaction to any components or excipients of the TIL therapy or the other study drugs: NMA-LD (cyclophosphamide, mesna, and fludarabine); IL-2; any component of the TIL infusion product formulation including human serum albumin (HSA), IL-2, and dextran-40
* Any other condition that in the investigator's judgement would significantly increase the risks of participation
* Patient has any complication or delayed healing from excisional procedure that in the investigator's opinion would increase the risks of lymphodepletion, adoptive TIL therapy and adjuvant IL-2
* Patients has a decline in performance status to ECOG > 1 (at the visit prior to admission for lymphodepletion)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Jazaeri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Amaria R, Knisely A, Vining D, Kopetz S, Overman MJ, Javle M, Antonoff MB, Tzeng CD, Wolff RA, Pant S, Lito K, Rangel K, Fellman B, Yuan Y, Lu KH, Sakellariou-Thompson D, Haymaker CL, Forget MA, Hwu P, Bernatchez C, Jazaeri AA. Efficacy and safety of autologous tumor-infiltrating lymphocytes in recurrent or refractory ovarian cancer, colorectal cancer, and pancreatic ductal adenocarcinoma. J Immunother Cancer. 2024 Feb 2;12(2):e006822. doi: 10.1136/jitc-2023-006822. PMID 38309721
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 08/17/2018 and the first participant was registered on study 10/16/2018. The study was closed to new patient entry on 04/02/2021 and the study was completed on 08/21/2024. All recruitments were done in a medical clinic setting.
Groups:
- Autologous TIL: Lymphodepletion therapy followed by autologous expanded TIL infusion then high dose IL-2 infusion
Period: Overall Study
Arm/Group | Autologous TIL
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Autologous TIL
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 54.4 [33 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Participants With Ovarian Cancer (OVCA), PDAC (Pancreatic Cancer), and Colorectal Cancers (CRC) According to RECIST v1.1 in Subjects With Ovarian Cancer (OVCA), PDAC (Pancreatic Cancer), and Colorectal Cancers (CRC)
Description: The ORR is derived as the sum of the number of patients with a confirmed CR or partial response (PR) divided by the number of patients in the All-Treated analysis set x 100%.
Time Frame: Through 4 years
Measure: Number (97.5% Confidence Interval); unit: Precentage of Participants
Arm/Group | Autologous TIL
Number analyzed (Participants) | 16
Precentage of Participants | 0 [0 to 21]

2. Secondary Outcome: Number of Participants With Stable Disease
Description: Participants will be evaluated at 6 and 12 weeks for response.
Time Frame: 6 weeks, 12 weeks
Measure: Number; unit: participants
Arm/Group | Autologous TIL
Number analyzed (Participants) | 16
participants
  Stable Disease at 6 weeks | 10
  Stable Disease at 12 weeks | 5

3. Secondary Outcome: Progression-free Survival (PFS) and Overall Survival (OS)
Time Frame: 44.8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Autologous TIL
Number analyzed (Participants) | 16
months
  PFS | 2.53 [1.54 to 4.11]
  OS | 18.86 [4.86 to NA] — Not reached.

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Autologous TIL
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous TIL (N=16)
Hepatobiliary disorder - drug induced liver toxicity (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous TIL (N=16)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 9 (11)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 14 (15)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CPK increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Edema limbs (General disorders) | 6 (6)
Edema trunk (General disorders) | 2 (2)
Fatigue (General disorders) | 14 (20)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 6 (6)
Flushing (Vascular disorders) | 3 (3)
General disorders - fluid overload (General disorders) | 4 (4)
General disorders - fluid retention (General disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (6)
Hot flashes (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (12)
Neutrophil count decreased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 13 (18)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 6 (6)
Skin disorder - other, macular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder - other, erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders - Other, fluid overload (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Weight gain (Investigations) | 6 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT03610490/Prot_SAP_000.pdf